CLINICAL TRIAL: NCT03651024
Title: A Prospective, First in Human Study to Evaluate the Safety and Performance of a Flow Modification System
Brief Title: Sano V First In Human Study to Treat ED
Acronym: FMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sano V Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN0001
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Erectile Dysfunction (ED)
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treating Patients with ED (Other): Treatment of patients with ED
  Interventions: Device: ED surgery

INTERVENTIONS:
Device: ED surgery — The surgical implant for ED treatment

SUMMARY:
A Prospective, First in Human Study to Evaluate the Safety and Performance of a Flow Modification System

ELIGIBILITY:
Inclusion Criteria:

1. Patient understands and has signed the study informed consent form.
2. Documented history of erectile dysfunction
3. Sexually active

Exclusion Criteria:

- 1. Current participation in any clinical study with any investigational drug or device.

2. Patient is known or suspected not to tolerate the procedure, including exposure to contrast 3. Active infection or fever that may be due to infection 4. Life expectancy < 2 years due to other illnesses

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 10 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
The surgical implant for ED treatment | 12 months
  Primary Safety Endpoint
  • 30-day Freedom from Major Adverse Events